CLINICAL TRIAL: NCT06976697
Title: Safety And Efficacy of Remotely Supervised Home-Based tDCS Treatment Of Major Depressive Disorder
Brief Title: Home-Based tDCS Treatment Of Major Depressive Disorder
Acronym: REACH-tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sooma Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM-001
Record Dates: First submitted 2025-05-07; First posted 2025-05-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Depression; Brain stimulation; Brain; Sooma; tDCS; tES
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active treatment (Experimental)
  Interventions: Device: Transcranial direct current stimulation
- Sham treatment (Sham Comparator)
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — In tDCS treatment session electrical current (2 mA) is applied for 30 minutes through two electrodes placed on top of scalp to modulate neural activity.
  Arms: Active treatment
Device: Sham transcranial direct current stimulation — Sham treatment mimics the active device use and the experiences from the active stimulation while minimizing active effects.
  Arms: Sham treatment

SUMMARY:
The REACH-tDCS study will evaluate the safety and efficacy of a noninvasive, at-home self-administered Sooma tDCS brain stimulation treatment for Major Depressive Disorder. The study uses randomized, blinded, placebo controlled design. The participants are assessed with video interviews and self-reports during the study, which lasts for 10 weeks followed by an optional continuation period.

DETAILED DESCRIPTION:
The study stages include: screening, eligibility evaluation, randomization to active or sham arm (1:1), the first treatment period (weeks 1-10) with sham-control and the optional open-label phase (weeks 11-20) where all treatments will be in active mode.

ELIGIBILITY:
Inclusion Criteria:

* 22 - 70 years of age
* Diagnosis of Unipolar MDD (DSM-V)
* PHQ-9 score of ≥13 AND MADRS score of ≥ 20 at baseline
* Antidepressant medication ongoing
* If in psychotherapy, have maintained stable psychotherapy
* Have access to a smartphone or other device running Android 7.0+ or iPhone Operating System (iOS) 13+
* Be under the care of a psychiatrist or a primary care physician
* Allow communication between the investigators/study staff and any healthcare provider who currently provides and/or has provided service to the patient/subject within at least two years
* Provide the name and contact of at least two adult persons who reside within a 60-minute drive of the patient's residence.
* Be able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study
* Be willing and able to comply with all study procedures
* Agree to meet all of the inclusion criteria throughout their participation in the study. Otherwise, the subject will be discontinued from the study
* Be able to understand, speak, and read English sufficient for the completion of trial assessments

Exclusion Criteria:

* Current state of mania or psychosis, or have a history of mania or psychosis.
* Treatment resistant depression.
* Are diagnosed with vitamin or hormonal deficiencies that may mimic mood disorders, as determined by the investigator.
* Be currently receiving any other interventional therapy for MDD other than a stable regimen of antidepressants or psychotherapy as defined in the inclusion criteria or have a history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), cranial electrotherapy stimulation (CES), transcranial direct current stimulation (tDCS), deep brain stimulation (DBS), or other brain stimulation.
* Have moderate or greater suicidality risk, or an attempt of suicide during lifetime or any previous hospitalization for suicidal behavior.
* Have sleep apnea (unless they are on CPAP treatment and are compliant with treatment) or a diagnosis of insomnia that is unrelated to depression, as determined by the investigator.
* Have any structural lesion or any neurocranial defect or any other clinically significant abnormality that might affect safety, study participation, or confound interpretation of study results, as determined by the investigator.
* Have any implant in the brain (e.g., DBS) or neurocranium, or any other active implantable medical device anywhere in the body (e.g. pacemaker, insulin pump).
* Have a history of epilepsy or seizures.
* Have shrapnel or any ferromagnetic material in the head.
* Have any disorder that would impair the ability to complete the study questionnaires.
* Have been diagnosed with autism spectrum disorder.
* Have an alcohol use disorder or substance use disorder (past 12 months).
* Have a cognitive impairment (including dementia).
* medications that affect cortical excitability, as determined by the investigator.
* Have ever taken esketamine / ketamine for treatment of depression.
* Are currently admitted or have ever been admitted to the hospital for depression.
* Have ever been diagnosed with obsessive-compulsive disorder (OCD) or bipolar type 1 or 2 disorder.
* Be diagnosed with PTSD, agoraphobia, anorexia or bulimia, panic or personality disorder, with active symptoms, based on the investigator's judgment.
* Have any history of myocardial infarction, coronary artery bypass graft (CABG), coronary heart failure (CHF), or history of other cardiac issues.
* Be currently experiencing or have a history of intractable migraines.
* Be a chronic tobacco smoker.
* Be currently pregnant or breastfeeding or planning to become pregnant or breastfeed any time during the study, or lack a medically acceptable method of contraception in females with child-bearing potential.
* Be currently incarcerated.
* Be participating concurrently in another clinical investigation or have participated in a clinical investigation within the last 90 days or intend to participate in another clinical investigation during the study.
* Have a hairstyle or hair type, such as very thick hair or voluminous hairstyle, that would prevent wearing of the treatment cap tightly enough on the head that the electrodes are held close to the scalp.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
MADRS: change from baseline | 10 weeks from treatment initiation.
  Mean change in depressive symptoms, measured by the Montgomery-Asberg Depression Rating Scale (MADRS) total score, from baseline to week 10. MADRS ranges from 0 to 60, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
MADRS: rate of response | 10 weeks from treatment initiation.
  Rate of response defined as the percent of subjects achieving at least 50% reduction from baseline in their MADRS at week 10.
MADRS: rate of remission | 10 weeks from treatment initiation.
  Rate of remission remission defined as the percent of subjects with MADRS score ≤ 10 at week 10.
HAM-D17: change form baseline | 10 weeks from treatment initiation.
  Mean change in depressive symptoms, measured by Hamilton Depression Rating Scale (17-items) (HAM-D17), from baseline to week 10. HAM-D17 ranges from 0 to 52, with higher scores indicating more severe depression.
HAM-D17: rate of response | 10 weeks from treatment initiation.
  Rate of response defined as the percent of subjects achieving at least 50% reduction from baseline in their HAM-D17 at week 10.
HAM-D17: rate of remission | 10 weeks from treatment initiation.
  Rate of remission defined as the percent of subjects with HAM-D17 score ≤ 7 at week 10.
PHQ-9: change from baseline | 10 weeks from treatment initiation.
  Mean change in depressive symptoms, measured by Patient Health Questionnaire-9 (PHQ-9) total score, from baseline to week 10. PHQ-9 ranges from 0 to 27, with higher scores indicating more severe depression.
PHQ-9: rate of response | 10 weeks from treatment initiation.
  Rate of response defined as the percent of subjects achieving at least 50% reduction from baseline in their PHQ-9 at week 10.
PHQ-9: rate of remission | 10 weeks from treatment initiation.
  Rate of remission, defined as the percent of subjects with PHQ-9 score ≤ 4 at week 10.
CGI-I | 10 weeks from treatment initiation.
  The clinical global impression - improvement scale (CGI-I) is a 7-point scale allowing the clinical rater to assess how much the patient's overall condition has improved or worsened since starting the intervention (1. very much improved, 2. much improved, 3. minimally improved, 4. no change, 5. minimally worse, 6. much worse, 7. very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Reist, M.D., Principal Investigator
Locations (1):
- Lindus Health (virtual study site), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD used in the results of the publication will be shared.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Beginning 1 year and ending 3 years after the publication of results.
Access Criteria: The deidentified IPD and the data dictionary will be provided for non-commercial use, via a data request, once an appropriate analysis plan has been provided and it has been approved by independent review and the study sponsor and a data sharing agreement has been signed. Data sharing will abide by the rules and policies defined by the sponsor, and relevant institutional review boards, as well as local, state and federal laws and regulations. Rights and privacy of individuals participating in the research will be protected at all times.

REFERENCES:
- See also: More information on this trial can be found on the Study Website. — https://www.lindushealth.com/research/reach-tdcs